CLINICAL TRIAL: NCT04918693
Title: A Study to Evaluate the Performance and Potential Benefits of an Assistive Artificial Intelligence Device ScanNav Anatomy Peripheral Nerve Block - US V1.0 for Ultrasound-guided Regional Anesthesia
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2021_AG_08
Record Dates: First submitted 2021-05-25; First posted 2021-06-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2021-06

CONDITIONS: Ultrasound Imaging of Anatomical Structures
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Participant: All 15 participants must be anesthesiologists who are competent to perform UGRA independently. In order to be eligible for the study, participants must be a U.S. board-eligible/board-certified and licensed Medical Doctor.
  Interventions: Device: Ultrasound scanning
- Trainee: All 15 trainees must be healthcare practitioners who are licensed to perform UGRA. In order to be eligible for the study, participants must be a U.S. board-eligible/board-certified health practitioner
  Interventions: Device: Ultrasound scanning

INTERVENTIONS:
Device: Ultrasound scanning — All participants will scan with and without device and trainee on 4 models. The order of the device assistance and models will be randomized between participants, but participant will always have exposure to device first before supervising the trainee.

SUMMARY:
This is a single-center, prospective study to be undertaken at University of Oregon, Portland, USA. The aim is to provide data on the clinical performance of ScanNav Anatomy PNB for identification of anatomical structures during UGRA scanning, in particular:

1. Assess the benefits of the device to intended users when supervising a trainee who is performing UGRA scanning.
2. Assess the benefits of the device when intended users perform UGRA scanning.
3. Assess risk mitigation by the intended users when performing UGRA scanning.

DETAILED DESCRIPTION:
Background:

The American Society of Regional Anesthesia and Pain Medicine (ASRA) has published evidence-based assessment of ultrasound-guided regional anesthesia (Neal et al., 2010) concluding that ultrasound guidance is superior or equal to other non-ultrasound nerve localization techniques. A subsequent publication from ASRA (Neal et al., 2016), has strengthened their position of ultrasound guidance being superior than other methods, including for the reduction of local anesthetic systemic toxicity. However, ultrasound-guided regional anesthesia (UGRA) is a difficult technique to master. A key activity of UGRA is ultrasound image interpretation (Sites et al., 2009) which ScanNav Anatomy PNB is designed to support.

Methodology:

15 participants (anesthesiologists capable of independently performing UGRA) will be recruited to evaluate the performance and benefit of ScanNav Anatomy PNB device in person, by scanning 2 healthy models (n=1 BMI<30, n=1 BMI>=30 kg/m2).

The device performance and benefits will be ascertained once the scanning session for each block is complete by use of a structured questionnaire.

* Participants will be asked to scan a model with and without the use of ScanNav Anatomy PNB. The order of with/without the device will be randomized between participants.
* Participants will also be asked to supervise a trainee (another healthcare professional qualified to perform the UGRA procedure under supervision) while they are scanning models with and without ScanNav Anatomy PNB aid. The participant will always use the device first before supervising the trainee.
* The above will be performed on 2 models from different BMI categories (n=1 BMI<30, n=1 BMI>=30 kg/m2; total scans n=16).
* The order of models will be randomized between participants.
* All 9 supported regions will be evaluated; each region will be scanned/evaluated at least 3 times.

Data collection

- Participants and trainees will be asked to complete a structured questionnaire to assess the device performance and clinical benefits at the end of scanning for the block.

Data analysis:

* Data will be aggregated and evaluated on safety critical structure type basis.
* Quantitative data obtained from the participants will be presented as frequencies and expressed as percent of total or as mean ± s.d. where appropriate.

The collected data and overall performance and benefits of ScanNav Anatomy PNB will be evaluated and summarized by presence and absence of ScanNav Anatomy PNB assistance, trainee and stratified by low/high BMI model.

Independent expert evaluation

* The scans be recorded during the study sessions. These scans will be post processed to short clips (10 seconds prior to obtaining optimum view) and sent for evaluation to an independent expert panel.
* The expert panel will be asked to evaluate the scans and the ScanNav Anatomy PNB highlighting performance independently from the participant. The majority opinion (at least 2/3) will be obtained to establish the agreement (e.g., yes/yes/no = yes)
* The answers obtained during the scan session from participants will be compared to expert panel view. Independent comparisons between performance assessment will be made, providing that the expert panel view is the 'ground truth'.
* Data will be evaluated and presented by safety structure on each model and overall (i.e., total for each class of safety critical structure; nerve, artery etc.).

ELIGIBILITY:
Participant Inclusion criteria

1. Completed advanced training (e.g., fellowship) in or hold a qualification related to UGRA
2. Regularly delivers direct clinical care using UGRA, including for 'awake' surgery where indicated
3. Member of a relevant professional society (e.g., ASA, ASRA, ESRA, RA-UK)
4. Regularly teach UGRA in the course of their clinical work, including advanced techniques where indicated

Participant exclusion criteria

1. Unwilling or unable to provide informed consent.
2. Involved in development of the ScanNav Anatomy PNB device.

Trainee Inclusion criteria

1. U.S. board-eligible/board-certified health practitioner who holds a qualification licensing to perform UGRA
2. NOT capable or confident of independent UGRA practice

Trainee exclusion criteria

1. Unwilling or unable to provide informed consent.
2. Involved in development of the ScanNav Anatomy PNB device.

Models Inclusion Criteria

1. Male or female, at least 18 years of age;
2. Able to comprehend and sign the Informed Consent prior to enrolment in the study.
3. To fit either BMI category: BMI <30 OR BMI >=30

Model Exclusion Criteria

1. Aged <18 years of age or over 60 years or age
2. Unwilling or unable to provide informed consent.
3. BMI> 39 kg/m2
4. Known pathology of the area to be scanned.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants All participants must be anesthesiologists who are competent to perform UGRA independently. In order to be eligible for the study, participants must be a U.S. board-eligible/board-certified and licensed Medical Doctor.
  Trainees All trainees must be healthcare practitioners who are licensed to perform UGRA. In order to be eligible for the study, participants must be a U.S. board-eligible/board-certified health practitioner.
  Models 4 models will be selected carefully based on their BMI inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-05-16 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Obtaining the correct ultrasound view | 6 months
  Number of participants obtaining the correct ultrasound view [majority view, at least 8/15 participants in agreement]

SECONDARY OUTCOMES:
Identifying anatomical structures | 6 months
  Number of participants identifying the correct anatomical structures in adult patients up to BMI 35 kg/m2 [majority view, at least 8/15 participants in agreement]
Effect of supervision in anatomical structure identification | 6 months
  Number of participants identifying the correct anatomical structures while being supervised in UGRA scanning [majority view, at least 8/15 participants in agreement]
Measuring operator confidence | 6 months
  Number of participants with improved confidence [majority view, at least 8/15 participants in agreement]
Number of errors in anatomy recognition by participants | 6 months
  Number of errors in anatomy recognition by participants [per class of safety critical structure, for all models]

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Woodworth, MD, Principal Investigator — Oregon Health and Science University; James Bowness, MD, Principal Investigator — University of Oxford & Royal Gwent Hospital
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bowness JS, El-Boghdadly K, Woodworth G, Noble JA, Higham H, Burckett-St Laurent D. Exploring the utility of assistive artificial intelligence for ultrasound scanning in regional anesthesia. Reg Anesth Pain Med. 2022 Jun;47(6):375-379. doi: 10.1136/rapm-2021-103368. Epub 2022 Jan 28. PMID 35091395